CLINICAL TRIAL: NCT04380142
Title: A Randomized, Double-Blind, Double-Dummy, Active-Controlled Study Comparing the Efficacy, Safety and Tolerability of ABBV-951 to Oral Carbidopa/Levodopa in Advanced Parkinson's Disease Patients
Brief Title: Study Comparing Continuous Subcutaneous Infusion Of ABBV-951 With Oral Carbidopa/Levodopa Tablets For Treatment Of Motor Fluctuations In Adult Participants With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-736; 2019-003930-18 (EudraCT Number)
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease (PD); ABBV-951; Levodopa/Carbidopa (LD/CD); Levodopa Phosphate/Carbidopa Phosphate (LDP/CDP)
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABBV-951 + Placebo for Levodopa/Carbidopa (LD/CD) (Experimental): After an open-label LD/CD Stabilization Period, participants will receive double-blind ABBV-951 by continuous subcutaneous infusion (CSCI) and oral placebo for LD/CD for 12 weeks
  Interventions: Drug: ABBV-951; Drug: Placebo for Levodopa/Carbidopa (LD/CD)
- Levodopa/Carbidopa (LD/CD) + Placebo for ABBV-951 (Active Comparator): After an open-label LD/CD Stabilization Period, participants will receive double-blind oral LD/CD and CSCI of placebo for ABBV-951 for 12 weeks
  Interventions: Drug: Levodopa/Carbidopa (LD/CD); Drug: Placebo for ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — Solution for continuous subcutaneous infusion (CSCI)
  Arms: ABBV-951 + Placebo for Levodopa/Carbidopa (LD/CD)
Drug: Placebo for Levodopa/Carbidopa (LD/CD) — Oral capsule
  Arms: ABBV-951 + Placebo for Levodopa/Carbidopa (LD/CD)
Drug: Levodopa/Carbidopa (LD/CD) — Oral encapsulated tablet
  Arms: Levodopa/Carbidopa (LD/CD) + Placebo for ABBV-951
Drug: Placebo for ABBV-951 — Solution for continuous subcutaneous infusion (CSCI)
  Arms: Levodopa/Carbidopa (LD/CD) + Placebo for ABBV-951

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study measures the efficacy, safety, and tolerability of ABBV-951 versus oral Levodopa (LD)/Carbidopa (CD) [LD/CD] in advanced PD participants to achieve reduction in motor fluctuations.

ABBV-951 is an investigational (unapproved) drug containing Levodopa Phosphate/Carbidopa Phosphate (LDP/CDP) given subcutaneously (under the skin) for the treatment of Parkinson's Disease. Adult participants with advanced PD will be enrolled. Approximately 130 participants will be enrolled in the study in approximately 80 sites across the world.

In one arm, participants will receive ABBV-951 solution as a continuous infusion under the skin plus oral placebo capsules for LD/CD. In the second arm, participants will receive placebo solution for ABBV-951 as a continuous infusion under the skin plus oral capsules containing LD/CD tablets. The treatment duration is 12 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease (PD) that is levodopa-responsive.
* Participant must be taking a minimum of 400 milligrams/day (mg/day) of Levodopa (LD) equivalents and be judged by the investigator to have motor symptoms inadequately controlled by current therapy, have a recognizable/identifiable "Off" and "On" states (motor fluctuations), and have an average "Off" time of at least 2.5 hours/day over 3 consecutive PD Diary days with a minimum of 2 hours each day.
* Participant or caregiver, if applicable, demonstrates the understanding and correct use of the delivery system, including the insertion of the cannula into the participant's abdomen, as assessed by the investigator or designee during the Screening period.

Exclusion Criteria:

* Clinically significant, unstable medical conditions or any other reason that the investigator determines would interfere with the participant's participation in this study or would make the participant an unsuitable candidate to receive study drug.
* History of allergic reaction or significant sensitivity to LD or constituents of the study drug (and its excipients) and/or other products in the same class.
* Participant has not received deep brain stimulation, CD/LD enteral suspension, or any other PD medication as continuous daily infusion, whether commercially available or investigational. Previous exposure to ABBV-951 is not allowed.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (76):
- United States (70):
  - University of Alabama at Birmingham - Main /ID# 216595, Birmingham, Alabama
  - University of South Alabama /ID# 216757, Mobile, Alabama
  - Xenoscience, Inc /ID# 217110, Phoenix, Arizona
  - Barrow Neurological Institute /ID# 216566, Phoenix, Arizona
  - HonorHealth /ID# 216642, Phoenix, Arizona
  - Movement Disorders Center of Arizona /ID# 216503, Scottsdale, Arizona
  - Banner Sun Health Res Inst /ID# 216507, Sun City, Arizona
  - University of Arkansas for Medical Sciences /ID# 216501, Little Rock, Arkansas
  - The Parkinson's & Movement Disorder Institute - Fountain Valley /ID# 216705, Fountain Valley, California
  - Neuro Pain Medical Center /ID# 216551, Fresno, California
  - University of California, San /ID# 216598, La Jolla, California
  - Loma Linda University Medical /ID# 216500, Loma Linda, California
  - Collaborative Neuroscience Research - Long Beach /ID# 216970, Long Beach, California
  - University of California, Los Angeles /ID# 216674, Los Angeles, California
  - SC3 Research Group - Pasadena /ID# 216821, Pasadena, California
  - Cedars-Sinai Medical Center-West Hollywood /ID# 216561, West Hollywood, California
  - University of Colorado Hospital /ID# 216527, Aurora, Colorado
  - Alpine Clinical Research Center /ID# 216637, Boulder, Colorado
  - Denver Neurological Research, LLC /ID# 216784, Denver, Colorado
  - Rocky Mountain Movement Disorders Center /ID# 216737, Englewood, Colorado
  - Christiana Care Health Service /ID# 216515, Newark, Delaware
  - Georgetown University Hospital /ID# 216632, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton /ID# 216517, Boca Raton, Florida
  - Brain Matters Research /ID# 217089, Delray Beach, Florida
  - Fixel Institute for Neurological Diseases /ID# 216514, Gainesville, Florida
  - Visionary Investigators Network - Miami /ID# 216679, Miami, Florida
  - Renstar Medical Research /ID# 216765, Ocala, Florida
  - Neurology Associates Ormond Beach /ID# 216521, Ormond Beach, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida /ID# 222656, Port Charlotte, Florida
  - University of South Florida /ID# 216638, Tampa, Florida
  - Premiere Research Institute - Palm Beach /ID# 217207, West Palm Beach, Florida
  - Duplicate_Atlanta Center for Medical Res /ID# 217091, Atlanta, Georgia
  - The Neurological Center of North Georgia /ID# 216499, Gainesville, Georgia
  - Rush University Medical Center /ID# 216567, Chicago, Illinois
  - University of Chicago Medical /ID# 217187, Chicago, Illinois
  - Indiana Clinical Research Cent /ID# 216615, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 216528, Kansas City, Kansas
  - St Elizabeth's Medical Center - Brighton /ID# 216716, Brighton, Massachusetts
  - Michigan State University /ID# 217158, East Lansing, Michigan
  - Clinical Research Professionals - Chesterfield /ID# 216669, Chesterfield, Missouri
  - St. Luke's Hosp. of Kansas City /ID# 216633, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 216548, St Louis, Missouri
  - Global Neurosciences Institute /ID# 217875, Lawrenceville, New Jersey
  - Northwell Health /ID# 216833, Lake Success, New York
  - Mount Sinai Beth Israel /ID# 216712, New York, New York
  - University of Rochester /ID# 218737, Rochester, New York
  - Wake Forest Univ HS /ID# 216522, Winston-Salem, North Carolina
  - Ohio State University - Wexner Medical Center /ID# 216900, Columbus, Ohio
  - The Orthopedic Foundation /ID# 217157, New Albany, Ohio
  - The Movement Disorder Clinic of Oklahoma /ID# 216860, Tulsa, Oklahoma
  - Legacy Research Institute /ID# 216558, Portland, Oregon
  - University of Pennsylvania /ID# 216560, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital /ID# 216553, Philadelphia, Pennsylvania
  - Prisma Health-Upstate /ID# 216594, Greenville, South Carolina
  - Premier Neurology, P.C. /ID# 217308, Greer, South Carolina
  - Coastal Neurology /ID# 217190, Port Royal, South Carolina
  - KCA Neurology - Franklin /ID# 217419, Franklin, Tennessee
  - Vanderbilt University Medical Center /ID# 216675, Nashville, Tennessee
  - Houston Pulmonary Sleep and Allergy Associates /ID# 216942, Cypress, Texas
  - Kerwin Research Center /ID# 216587, Dallas, Texas
  - Neurology Consultants of Dallas - LBJ Fwy /ID# 216564, Dallas, Texas
  - Texas Movement Disorder Specialists /ID# 216523, Georgetown, Texas
  - Houston Methodist Hospital /ID# 216707, Houston, Texas
  - Central Texas Neurology Consul /ID# 216629, Round Rock, Texas
  - University of Utah Health Care /ID# 216710, Salt Lake City, Utah
  - Meridian Clinical Research /ID# 216731, Norfolk, Virginia
  - Neurological Associates - Forest Ave /ID# 216636, Richmond, Virginia
  - Swedish Neuroscience /ID# 216526, Seattle, Washington
  - Inland Northwest Research /ID# 221036, Spokane, Washington
  - Medical College of Wisconsin /ID# 216498, Milwaukee, Wisconsin
- Australia (6):
  - Liverpool Hospital /ID# 218681, Liverpool, New South Wales
  - Westmead Hospital /ID# 216535, Westmead, New South Wales
  - Gold coast University Hospital /ID# 218373, Southport, Queensland
  - Royal Adelaide Hospital /ID# 216533, Adelaide, South Australia
  - Kingston Centre /ID# 216537, Cheltenham, Victoria
  - The Royal Melbourne Hospital /ID# 216536, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Antonini A, Bergmans B, Kern DS, Gandor F, Nishikawa N, Standaert DG, Fritz B, Gupta R, Nozaki T, Shah MB, Bergmann L, Kimber T. Foslevodopa/Foscarbidopa in Younger Patients Earlier Within Advanced Parkinson's Disease: Post Hoc Analysis of a Randomized Trial. Neurol Ther. 2026 Feb;15(1):309-324. doi: 10.1007/s40120-025-00856-1. Epub 2025 Dec 1. PMID 41324738
- [Derived] Pahwa R, Aldred J, Soileau MJ, Standaert DG, Fung VSC, Kimber T, Malaty IA, Santos-Garcia D, Carroll C, Henriksen T, Parab A, Yan CH, Facheris MF, Spiegel A, Harmer L, Zamudio J, Chaudhuri KR. Improvement in Motor Consistency and Stability with Foslevodopa/Foscarbidopa in Advanced Parkinson's Disease: Post Hoc Analysis of Two Phase 3 Clinical Trials. Neurol Ther. 2025 Dec;14(6):2491-2506. doi: 10.1007/s40120-025-00827-6. Epub 2025 Oct 4. PMID 41045349
- [Derived] Soileau MJ, Aldred J, Budur K, Fisseha N, Fung VS, Jeong A, Kimber TE, Klos K, Litvan I, O'Neill D, Robieson WZ, Spindler MA, Standaert DG, Talapala S, Vaou EO, Zheng H, Facheris MF, Hauser RA. Safety and efficacy of continuous subcutaneous foslevodopa-foscarbidopa in patients with advanced Parkinson's disease: a randomised, double-blind, active-controlled, phase 3 trial. Lancet Neurol. 2022 Dec;21(12):1099-1109. doi: 10.1016/S1474-4422(22)00400-8. PMID 36402160

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants entered an open-label oral Levodopa/Carbidopa (LD/CD) Stabilization Period of 14 to 21 days, at the end of which, eligible participants were randomized 1:1 to 12 weeks of treatment with either: 24-hour/day continuous subcutaneous infusion (CSCI) of ABBV-951 + oral placebo capsules for LD/CD immediate-release (IR) or 24-hour/day CSCI of placebo solution for ABBV-951 + encapsulated LD/CD IR tablets in a 12-week Double-Blind Treatment Period.
Groups:
- LD/CD Stabilization Period: The dose and schedule of oral LD/CD were adjusted over the first 7 to 14 days by the investigator to achieve the best possible control of the participant's motor symptoms; that included using nighttime dosing if needed and was agreed upon by the participant and the investigator. Once stabilized, no further adjustments to oral LD/CD IR were to be made for at least 7 days prior to randomization.
- LD/CD + Placebo for ABBV-951: Participants received oral LD/CD and CSCI of placebo for ABBV-951 for 12 weeks.
- ABBV-951 + Placebo for LD/CD: Participants received ABBV-951 by CSCI and oral placebo for LD/CD for 12 weeks.
Period: LD/CD Stabilization Period
Arm/Group | LD/CD Stabilization Period | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Started | 174 | 0 | 0
Completed | 145 | 0 | 0
Not Completed | 29 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Difficulty With Drug Delivery System | 2 | 0 | 0
Not completed — Other, Not Specified | 18 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | LD/CD Stabilization Period | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Started (Number Randomized) | 0 | 69 | 76
Randomized and Treated | 0 | 67 | 74
Completed | 0 | 62 | 48
Not Completed | 0 | 7 | 28
Not completed — Adverse Event | 0 | 1 | 14
Not completed — Withdrew Consent | 0 | 3 | 6
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Difficulty With Drug Delivery System | 0 | 1 | 3
Not completed — Other, Not Specified | 0 | 0 | 1
Not completed — Did Not Receive Study Drug | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received any dose of study drug during the Double-Blind Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD | Total
Number analyzed (Participants) | 67 | 74 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.82) | 66.3 (9.20) | 66.4 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 24 | 42
  Male | 49 | 50 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 66 | 70 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 2 | 4
  White | 61 | 70 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Averaged Normalized On Time Without Troublesome Dyskinesia [Mean (Standard Deviation); unit: normalized hours] — "On" time without dyskinesia plus "On" time with non-troublesome dyskinesia are based on the Parkinson's Disease (PD) Diary (normalized to a 16-hour waking day averaged over 3 consecutive days). Baseline value is defined as the average of normalized "On" time without troublesome dyskinesia collected over the 3 PD Diary days before randomization. Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment.
  normalized hours
    number analyzed (Participants) | 67 | 73 | 140
    (all) | 9.49 (2.619) | 9.20 (2.423) | 9.34 (2.514)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Average Daily Normalized "On" Time Without Troublesome Dyskinesia
Description: "On" time is defined as periods of good motor symptom control, and was assessed by the Parkinson's Disease (PD) diary. The normalized "On" time without troublesome dyskinesia is the sum of the normalized "On" time without dyskinesia and the normalized "On" time with non-troublesome dyskinesia. "On" time without dyskinesia plus "On" time with non-troublesome dyskinesia are based on the PD Diary (normalized to a 16-hour waking day averaged over 3 consecutive days). Baseline value is defined as the average of normalized "On" time without troublesome dyskinesia collected over the 3 PD Diary days before randomization.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with a baseline and Week 12 assessment.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 62 | 47
hours | 0.97 (0.50) | 2.72 (0.52)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.0083, mixed model repeated measures — The model included fixed categorical effects of treatment, country and visit, baseline-by-visit and treatment-by-visit interactions, and baseline as a covariate. An unstructured variance-covariance matrix was used; Least Squares (LS) Mean of Difference = 1.75, 95% CI 2-sided [0.46 to 3.05], Standard Error of Mean 0.65

2. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Average Daily Normalized "Off" Time (Hours)
Description: "Off" time is defined as periods of poor mobility, tremor, slowness, and stiffness and was assessed by the PD Diary.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 62 | 47
hours | -0.96 (0.49) | -2.75 (0.50)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.0054, mixed model repeated measures — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.79, 95% CI 2-sided [-3.03 to -0.54], Standard Error of Mean 0.63

3. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II Score
Description: The Part II MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of PD. MDS-UPDRS is multimodal scale assessing impairment and disability. Part II assesses the participant's motor experiences of daily living with 13 questions. (The numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe). Part II scores range from 0 to 52, with higher scores indicating more severe symptoms of PD.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 62 | 46
score on a scale | -1.06 (0.79) | -2.65 (0.82)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.1318, mixed model repeated measures — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.58, 95% CI 2-sided [-3.65 to 0.48], Standard Error of Mean 1.05

4. Secondary Outcome: Early Morning "Off" Status (Morning Akinesia) at Week 12 of the Double-Blind Treatment Period
Description: Early morning "Off" status is assessed by the PD Diary as percentage of participants with early morning "Off" upon waking up at Week 12, based on the first morning symptom upon awakening on the last valid PD Diary day at Week 12.
  "Off" time is defined as periods of poor mobility, tremor, slowness, and stiffness and was assessed by the PD Diary.
Time Frame: Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with an assessment for morning akinesia at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 60 | 47
percentage of participants | 63.3 | 17.0
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p <= 0.001, generalized linear mixed model — The generalized linear mixed model: status = treatment country visit baseline treatment*visit. The unstructured variance-covariance structure is used; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.04 to 0.31], Standard Error of Mean 0.49

5. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Average Daily Normalized "On" Time Without Dyskinesia (Hours)
Description: "On" time is defined as periods of good motor symptom control, and was assessed by the PD diary. The normalized "On" time without dyskinesia is defined as the hours of average daily normalized "On" time without dyskinesia as assessed by the PD Diary (normalized to a 16-hour waking day averaged over 3 consecutive days).
  Baseline value is defined as the average of normalized "On" time without dyskinesia collected over the 3 PD Diary days before randomization.
Time Frame: Baseline, Week 12 of the double-blind treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 62 | 47
hours | 1.32 (0.53) | 3.13 (0.54)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.0091, generalized linear mixed model; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.46 to 3.16], Standard Error of Mean 0.68

6. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Parkinson's Disease Sleep Scale-2 (PDSS-2) Total Score
Description: The PDSS-2 addresses PD-specific sleep disturbances such as restless leg syndrome (RLS), morning akinesia, pain, and sleep apnea. The frequency is assessed for the 15 sleep problems based on a 5-point Likert-type scale (ranging from 0 [never] to 4 [very often]). Scores are calculated for each of the 3 domains (motor symptoms at night, PD symptoms at night, and disturbed sleep) as well as a total score. The PDSS-2 domain scores range from 0 to 20 and the total score is a sum of the 3 domains and ranges from 0 to 60. Higher scores indicate higher frequency and more severe impact of PD on sleep.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with an assessment for PDSS-2.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 44
score on a scale | -2.52 (1.12) | -7.92 (1.18)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p <= 0.001, ANCOVA — ANCOVA model including effects for treatment, country, and baseline; LS Mean of Difference = -5.40, 95% CI 2-sided [-8.03 to -2.78], Standard Error of Mean 1.32

7. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Quality of Life Assessed by Parkinson's Disease Questionnaire 39 Item (PDQ-39) Summary Index Score
Description: The PDQ-39 is a disease-specific instrument designed to measure aspects of health that are relevant to participants with PD, and which may not be included in general health status questionnaires. It evaluates the 8 dimensions of mobility, activities of daily living, emotional well-being, stigma, social support, cognition, and communication. Data from the PDQ-39 can be presented in either domain scores or as a summary index score. The full range of the PDQ-39 Summary Index score is from 0 (no patient-related symptoms/quality of life unaffected) to 100 (highest patient-related symptoms/low quality of life).
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with an assessment for PDQ-39.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 45
score on a scale | -2.28 (1.75) | -6.38 (1.83)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.0470, ANCOVA — ANCOVA model including effects for treatment, country, and baseline; Least Squares (LS) Mean of Difference = -4.10, 95% CI 2-sided [-8.14 to -0.05], Standard Error of Mean 2.04

8. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Quality of Life Assessed by the EuroQol 5-Dimension Questionnaire (EQ-5D-5L) Summary Index
Description: The EQ-5D-5L is a standardized non-disease specific instrument for describing and valuing health-related quality of life. The EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the subject's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. The health status is converted to an index value using the country-specific weighted scoring algorithm for the United States (US). The summary index value for the US ranges from a worst score of -0.109 to a best score of 1. An increase in the EQ-5D-5L total score indicates improvement.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with an assessment for EQ-5D-5L.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 44
score on a scale | 0.002 (0.021) | 0.051 (0.022)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.0566, ANCOVA — ANCOVA model including effects for treatment, country, and baseline; LS Mean of Difference = 0.049, 95% CI 2-sided [-0.001 to 0.100], Standard Error of Mean 0.025

9. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Median Bradykinesia Score (BK50) as Assessed by the Parkinson's KinetiGraph/Personal KinetiGraph (PKG) Wearable Device
Description: The PKG wearable device is an innovative mobile health technology that provides continuous, objective, ambulatory assessment of the symptoms of PD including tremor, bradykinesia, dyskinesia, and daytime somnolence. For each participant, the PKG watch collected data continuously and an algorithm calculated a bradykinesia score every 2 minutes between 9am-6pm across multiple days. Among these scores for this participant at this visit, the median of all the score values is defined as BK50. A higher score indicates worse bradykinesia (there is no prespecified range of scores). The BK50 scores for all participants across all visits were then analyzed with mixed-effect model for repeated measures (MMRM) and the LS mean (model-based mean) was obtained from the model.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with a baseline and Week 12 assessment for BK50 score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 66
score on a scale | -0.34 (0.52) | 1.38 (0.56)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.0184, Repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 1.72, 95% CI 2-sided [0.30 to 3.15], Standard Error of Mean 0.72

10. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Interquartile Range of Bradykinesia Score (BK75-BK25) as Assessed by the PKG Wearable Device
Description: The PKG wearable device is an innovative mobile health technology that provides continuous, objective, ambulatory assessment of the symptoms of PD including tremor, bradykinesia, dyskinesia, and daytime somnolence. For each participant, the PKG watch collected data continuously and an algorithm calculated a bradykinesia score every 2 minutes between 9am-6pm across multiple days. Among these scores for this participant at this visit, the median of all the score values is defined as BK50 (there is no prespecified range of scores). BK75-BK25 is the difference between the third quartile (BK75) and first quartile (BK25) bradykinesia scores, and this interquartile range is a measure of variability of bradykinesia. A higher score indicates a higher degree of variability in bradykinesia scores. The BK75 and BK 25 scores for all participants across all visits were then analyzed with mixed-effect model for repeated measures (MMRM) and the LS mean (model-based mean) was obtained from the model.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with a baseline and Week 12 assessment for BK75-BK25.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 66
score on a scale | 0.13 (0.49) | 0.31 (0.54)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.7989, Repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.18, 95% CI 2-sided [-1.20 to 1.55], Standard Error of Mean 0.69

11. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Median Dyskinesia Score (DK50) as Assessed by the PKG Wearable Device
Description: The PKG wearable device is an innovative mobile health technology that provides continuous, objective, ambulatory assessment of the symptoms of PD including tremor, bradykinesia, dyskinesia, and daytime somnolence. For each participant, the PKG watch collected data continuously and an algorithm calculated a dyskinesia score every 2 minutes between 9am-6pm across multiple days. Among these scores for this participant at this visit, the median of all the score values is defined as DK50. A higher score indicates worse dyskinesia (there is no prespecified range of scores). The DK50 scores for all participants across all visits were then analyzed with mixed-effect model for repeated measures (MMRM) and the LS mean (model-based mean) was obtained from the model.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with a baseline and Week 12 assessment for DK50.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 66
score on a scale | 1.02 (1.38) | -1.71 (1.41)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.1656, Repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -2.73, 95% CI 2-sided [-6.61 to 1.15], Standard Error of Mean 1.96

12. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Treatment Period in Interquartile Range of Dyskinesia Score (DK75-DK25) as Assessed by the PKG Wearable Device
Description: The PKG wearable device is an innovative mobile health technology that provides continuous, objective, ambulatory assessment of the symptoms of PD including tremor, bradykinesia, dyskinesia, and daytime somnolence. For each participant, the PKG watch collected data continuously and an algorithm calculated a dyskinesia score every 2 minutes between 9am-6pm across multiple days. Among these scores for this participant at this visit, the median of all the score values is defined as DK50 (there is no prespecified range of scores). DK75-DK25 is the difference between the third quartile (DK75) and first quartile (DK25) dyskinesia scores, and this interquartile range is a measure of variability of dyskinesia. A higher score indicates a higher degree of variability in dyskinesia scores. The DK75 and DK25 scores for all participants across all visits were then analyzed with mixed-effect model for repeated measures (MMRM) and the LS mean (model-based mean) was obtained from the model.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Full Analysis Set (FAS): all randomized participants who received any dose of study drug during the Double-Blind Treatment Period and who had baseline and at least 1 post-baseline observation for at least 1 efficacy assessment. Participants with a baseline and Week 12 assessment for DK75-DK25.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 59 | 66
score on a scale | 2.72 (2.59) | -2.77 (2.64)
Statistical Analysis 1: Comparison: LD/CD + Placebo for ABBV-951 vs ABBV-951 + Placebo for LD/CD; Test type: Superiority; p = 0.1347, Repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -5.49, 95% CI 2-sided [-12.71 to 1.73], Standard Error of Mean 3.65

13. Secondary Outcome: Number of Participants With Irritation Grade Numeric Grade >= 5 or Letter Grade >= D on the Infusion Site Irritation Scale Across All Study Post-Baseline Visits
Description: The investigator or qualified designee evaluated the infusion site area (abdomen). A 2-part (numeric and letter grading) evaluation scale was used to assess irritation. Irritation - Numeric Grades: 0 = No evidence of irritation; 1 = Minimal erythema, barely perceptible; 2 = Moderate erythema, readily visible; or minimal edema, or minimal papular response; 3 = Erythema and papules; 4 = Definite edema; 5 = Erythema, edema, and papules; 6 = Vesicular eruption; 7 = Strong reaction spreading beyond the test site. Irritation - Letter Grades: A = No finding; B = Slight glazed appearance; C = Marked glazing; D = Glazing with peeling and cracking; E = Glazing with fissures; F = Film of dried serous exudates covering all or portion of the patch site; G = Small petechial erosions and/or scabs.
Time Frame: Day 2 up to Week 12 of the double-blind treatment period plus 30 days
Population: Safety Analysis Set: participants who received any dose of study drug during the Double-Blind Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 67 | 74
Participants
  At Least 1 Observation of Numeric Grade >= 5 | 0 | 10
  At Least 1 Observation of Letter Grade >= D | 0 | 6
  At Least 1 Observation of Numeric Grade >= 5 or Letter Grade >= D | 0 | 10
  At Least 1 Observation of Numeric Grade >= 5 and Letter Grade >= D | 0 | 6

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) During the Oral LD/CD Stabilization Period
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with treatment. An AE, whether associated with study drug or not, meeting any of the following criteria is considered a serious AE (SAE): results in death; is life-threatening; results in hospitalization or prolongation of hospitalization; is a congenital anomaly; results in persistent or significant disability/incapacity; is an important medical event requiring medical or surgical intervention to prevent a serious outcome. The severity of each AE is rated as mild, moderate, or severe, and having either a reasonable possibility or no reasonable possibility of relationship to study drug. Events were considered treatment emergent if they arose after the first dose of study drug.
Time Frame: From first dose of stabilization period treatment up to the first dose of the double-blind treatment period
Population: Oral LD/CD Analysis Set: all participants who received at least 1 dose of open label CD/LD IR tablets during the Oral CD/LD Stabilization Period.
Measure: Count of Participants; unit: Participants
Arm/Group | LD/CD Stabilization Period
Number analyzed (Participants) | 174
Participants
  Any TEAE | 41
  Any Severe TEAE | 3
  Any TEAE Considered Related to Study Drug | 2
  Any TEAE Considered Associated With COVID-19 Infection | 0
  Any TEAE Leading to Premature Discontinuation of Study Drug | 3
  Any TEAE Leading Death | 0
  Any Serious TEAE | 4
  Deaths Related to COVID-19 | 0

15. Secondary Outcome: Number of Participants With TEAEs During the Double-Blind Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with treatment. An AE, whether associated with study drug or not, meeting any of the following criteria is considered an SAE: results in death; is life-threatening; results in hospitalization or prolongation of hospitalization; is a congenital anomaly; results in persistent or significant disability/incapacity; is an important medical event requiring medical or surgical intervention to prevent a serious outcome. The severity of each AE is rated as mild, moderate, or severe, and having either a reasonable possibility or no reasonable possibility of relationship to study drug. Adverse events of special interest include polyneuropathy, weight loss, somnolence, hallucinations/psychosis. Events were considered treatment emergent if they arose after the first dose of study drug.
Time Frame: From first dose of double-blind treatment up to Week 12 of the double-blind treatment period plus 30 days
Population: Safety Analysis Set: participants who received any dose of study drug during the Double-Blind Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 67 | 74
Participants
  Any TEAE | 42 | 63
  Any Serious TEAE | 4 | 6
  Any TEAE Leading to Death | 1 | 0
  Any TEAE Leading to Study Drug Discontinuation | 1 | 16
  Any Severe TEAE | 1 | 7
  Any TEAE Considered Related to Study Drug | 15 | 52
  Any Serious TEAE Considered Related With Infusion Pump | 0 | 3
  All Deaths (Includes Non-Treatment-Emergent Deaths) | 1 | 0
  Deaths Related to COVID-19 | 0 | 0
  Any Adverse Event of Special Interest | 25 | 59

16. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes From Baseline in Hematology, Chemistry, Urinalysis, Special Laboratory Parameters, Vital Signs, and Electrocardiograms (ECGs)
Description: Measures analyzed for prespecified potentially clinically significant criteria: hematology (hematocrit, hemoglobin, red blood cells, white blood cells, neutrophils, bands, lymphocytes, monocytes, basophils, eosinophils, platelets, mean corpuscular hemoglobin, mean corpuscular volume concentration, prothrombin time, activated partial thromboplastin time), laboratory (blood urea nitrogen, creatinine, creatine phosphokinase, bilirubin, alanine aminotransferase, aspartate aminotransferase, lactate dehydrogenase, gamma-glutamyl transpeptidase, alkaline phosphatase, sodium, potassium, calcium, phosphorus, uric acid, total protein, albumin, glucose, sodium bicarbonate, chloride, triglycerides, cholesterol, magnesium), special lab criteria (vitamin B12, vitamin B6, folate, homocysteine, methylmalonic acid), vital signs (diastolic and systolic blood pressure, pulse rate), ECG (heart rate, PR, and QTcF interval), urinalysis (specific gravity, ketones, pH, protein, glucose, blood, bilirubin).
Time Frame: Screening up to Week 12 of the double-blind treatment period
Population: Safety Analysis Set: participants who received any dose of study drug during the Double-Blind Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 67 | 74
Participants
  Hematology | 0 | 0
  Chemistry | 0 | 0
  Urinalysis | 0 | 0
  Special Laboratory Parameters | 0 | 0
  Vital Signs | 0 | 0
  ECGs | 0 | 0

17. Secondary Outcome: Number of Participants With Affirmative Responses on the Columbia-Suicide Severity Rating Scale (C-SSRS) Across All Study Post-Baseline Visits During the Double-Blind Treatment Period
Description: The C-SSRS is a systematically administered instrument developed to track suicidal adverse events across a treatment study. The instrument is designed to assess suicidal behavior and ideation, track and assess all suicidal events, as well as the lethality of attempts. Suicidal ideation categories include the following: wish to be dead; nonspecific active suicidal thoughts; active suicidal ideation without intent to act; active suicidal ideation with some intent to act but no plan; active suicidal ideation with plan and intent. Suicidal behavior categories include the following: actual attempt; interrupted attempt; aborted attempt; preparatory acts or behavior; suicidal behavior; completed suicide.
Time Frame: Screening up to Week 12 of the double-blind treatment period
Population: Safety Analysis Set: participants who received any dose of study drug during the Double-Blind Treatment Period. Participants with an assessment for C-SSRS.
Measure: Count of Participants; unit: Participants
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 67 | 74
Participants
  Participants With Any Suicidal Ideations | 2 | 5
  Participants With Any Suicidal Behaviors | 0 | 0
  Participants With Any Suicidal Behaviors or Ideations | 2 | 5
  Participants With Non-Suicidal Self-Injurious Behavior | 0 | 0

18. Secondary Outcome: Number of Participants With a Subscore > 5 For Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease - Ration Scale (QUIP-RS) at Any Time During the Double-Blind Treatment Period
Description: The QUIP-RS measures the severity of symptoms and support a diagnosis of impulse control disorders and related disorders in PD. QUIP-RS subscores include gambling (score 0 to 16), sex (score 0 to 16), buying (score 0 to 16), eating (score 0 to 16), hobbyism-punding (score 0 to 32), and PD medication use (score 0 to 16). Higher scores represent a worse outcome.
Time Frame: Baseline (Week 0) up to Week 12 of the double-blind treatment period
Population: Safety Analysis Set: participants who received any dose of study drug during the Double-Blind Treatment Period. Participants with at least 1 post-baseline value for the specific QUIP-RS subscore.
Measure: Count of Participants; unit: Participants
Arm/Group | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
Number analyzed (Participants) | 65 | 67
Participants
  Impulse Control Disorder: Buying Score | 3 | 3
  Impulse Control Disorder: Eating Score | 5 | 6
  Impulse Control Disorder: Gambling Score | 2 | 0
  Impulse Control Disorder: Sex Score | 6 | 4
  Additional Disorder: Hobbyism Punding Score | 12 | 7
  Additional Disorder: PD Medication Use Score | 5 | 6

ADVERSE EVENTS:
Time Frame: CD/LD Stabilization Period: From Screening (All-Cause Mortality) or first dose of stabilization period treatment (Serious/Other Adverse Events) up to the first dose of the double-blind treatment period. Double-Blind Treatment Period: From Screening (All-Cause Mortality) or first dose of double-blind treatment (Serious/Other Adverse Events) up to Week 12 of the double-blind treatment period plus 30 days.
Arm/Group | LD/CD Stabilization Period | LD/CD + Placebo for ABBV-951 | ABBV-951 + Placebo for LD/CD
All-Cause Mortality (participants affected / at risk) | 0/174 | 1/67 | 0/74
Serious Adverse Events (participants affected / at risk) | 4/174 | 4/67 | 6/74
Other Adverse Events (participants affected / at risk) | 15/174 | 18/67 | 51/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LD/CD Stabilization Period (N=174) | LD/CD + Placebo for ABBV-951 (N=67) | ABBV-951 + Placebo for LD/CD (N=74)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE HEPATITIS B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CATHETER SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFUSION SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PARKINSONISM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARKINSONISM HYPERPYREXIA SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DELUSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PARANOIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIAPHRAGM MUSCLE WEAKNESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LD/CD Stabilization Period (N=174) | LD/CD + Placebo for ABBV-951 (N=67) | ABBV-951 + Placebo for LD/CD (N=74)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
INFUSION SITE BRUISING (General disorders) | 1 (1) | 2 (2) | 6 (6)
INFUSION SITE ERYTHEMA (General disorders) | 0 (0) | 1 (1) | 20 (33)
INFUSION SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 6 (8)
INFUSION SITE INDURATION (General disorders) | 0 (0) | 0 (0) | 4 (5)
INFUSION SITE NODULE (General disorders) | 0 (0) | 0 (0) | 6 (8)
INFUSION SITE OEDEMA (General disorders) | 0 (0) | 0 (0) | 9 (15)
INFUSION SITE PAIN (General disorders) | 0 (0) | 1 (1) | 19 (29)
INFUSION SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 4 (5)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 4 (4)
INFUSION SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 13 (14)
INFUSION SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 6 (7) | 11 (14) | 6 (7)
BALANCE DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
DYSKINESIA (Nervous system disorders) | 5 (5) | 4 (4) | 8 (8)
ON AND OFF PHENOMENON (Nervous system disorders) | 2 (2) | 0 (0) | 6 (6)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (5)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04380142/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT04380142/SAP_001.pdf